CLINICAL TRIAL: NCT04227652
Title: Control of Fever in Septic Patients
Acronym: COVERSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KARIM-13-COVERSEP; RVO-FNOs/2013-2 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: sepsis; severe sepsis; septic shock; fever; ibuprofen; physiological reserves
MeSH Terms: conditions — Sepsis; Shock, Septic; Fever

STUDY DESIGN:
Intervention Model Description: The study subjects were enrolled in two parallel groups.
Masking Description: No masking was used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive treatment strategy (Experimental): The antipyretic strategy was initiated immediately upon increase of the temperature above 38.3°C. The antipyretic strategy consisted of administration of ibuprofen (per-orally or into the nasogastric tube, or rectal administration in the form of a suppository) in therapeutical dose, alway supplemented with physical cooling in cases when the temperature exceeded 39.5°C. The body temperature was measured in the urinary bladder.
  Interventions: Drug: Ibuprofen administration
- Conservative treatment strategy (Experimental): The antipyretic strategy was initiated only after the body temperature exceeded 39.5°C. The antipyretic strategy consisted of administration of ibuprofen (per-orally or into the nasogastric tube, or rectal administration in the form of a suppository) in therapeutical dose, alway supplemented with physical cooling in cases when the temperature exceeded 39.5°C. The body temperature was measured in the urinary bladder.
  Interventions: Drug: Ibuprofen administration

INTERVENTIONS:
Drug: Ibuprofen administration — Administration of ibuprofen, according to treatment recommendations - per orally, into the nasogastric tube, or in the form of a suppository

SUMMARY:
The benefits of fever treatment in critically ill patients remains unclear. The aim of the prospective, randomized clinical trial was to verify the hypothesis that the administration of ibuprofen in order to decrease the fever in septic patients without limited cardiorespiratory reserve leads to decreasing their prognosis.

DETAILED DESCRIPTION:
Fever is a frequently observed part of the organism's response to infection, and it is a well-known fact that it has positive effects, as it inhibits the growth of microorganisms, and potentiates the activity of anti-microbial agents. On the other hand, fever increases the demand of tissues for oxygen and increases the production of carbon dioxide in tissues. Adapting to these metabolic changes requires an efficient cardiorespiratory apparatus. In other words, in patients with a limited cardiorespiratory reserve (typically patients of higher age or patients with a serious disease of the heart or lungs), the beneficial anti-microbial effect of fever may be masked with cardiorespiratory maladaptation to fever-induced metabolic changes. Indeed, one of the randomized clinical trials investigating the effect of "aggressive" antipyretic strategy used in practice (administration of acetaminophen at the temperature > 38.5 degrees Celsius, and addition of physical cooling should the temperature exceed 39.5 degrees Celsius upon the prognosis of critically ill patients showed that the "aggressive" treatment of fever may result in higher mortality when compared with a "permissive" approach, i.e. an approach when the treatment of fever is initiated only after the body temperature has exceeded 40 degrees Celsius. The study differs remarkably from other studies performed among the population of critically ill patients, and also from studies, which did not manifest the effect of fever treatment upon the mortality of patients, with the age of patients. The average age of patients in both arms of the study was only 47 years of age, whereas the average age of patients in other studies was usually around 60 years of age. It is thus possible to presume that, due to the lower age, the patients in this study possessed a sufficient cardiorespiratory reserve for adaptation to metabolic changes induced with fever, which may have enabled a full manifestation of its anti-microbial effect, and may have led to better patient prognosis. The mortality rate in the group of patients with the "permissive" approach to fever treatment was only 2.6 percent, whereas, in the group of patients with the "aggressive" treatment, the mortality rate was 15.9 percent (p=0.06); due to this fact, the study was prematurely terminated by the Ethics Committee. Based on this study, we decided to test the hypothesis that the administration of ibuprofen in order to decrease the fever would lead to a worsening of the patient prognosis. Ibuprofen was selected due to its potent antipyretic effect, and also due to the fact that the favorable effect of its anti-inflammatory effect upon the prognosis of patients with sepsis has not been fully demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years of age
* body temperature >38.3°C within 2 consecutive hours
* anti-microbial therapy for a known or suspected infection

Exclusion Criteria:

* patients admitted after successful cardiopulmonary resuscitation (CPR)
* acute myocardial infarction
* brain injury (traumatic and non-traumatic)
* transfer from another ICU after 72 hours
* pregnancy
* antipyretic medication prior to randomization
* non-obtaining the informed consent
* moribund condition
* high risk of hemodynamic or respiratory maladaptation on the metabolic effect of fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
SOFA score value | up to 7 days
  The SOFA score (Sequential Organ Failure Assessment) was measured on Day 3 and Day 7

SECONDARY OUTCOMES:
Serum interleukin-6 level | up to 7 days
  The serum interleukin-6 level was measured on Day 3 and Day 7
Serum procalcitonine level | up to 7 days
  The serum procalcitonine level was measured on Day 3 and Day 7
Serum lactate level | up to 7 days
  The serum lactate level was measured on Day 3 and Day 7
Central venous oxygen saturation | up to 7 days
  The central venous oxygen saturation was measured on Day 3 and Day 7
Duration of artificial ventilation | 1 month
  The duration of artificial ventilation in days was observed
Duration of vasopressor support | 1 month
  The duration of vasopressor support in days was observed
Length of ICU stay | 1 month
  The length of ICU stay in days was observed
Length of hospital stay | 3 months
  The length of hospital stay in days was observed

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kula, MD,CSc., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There exists no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Schulman CI, Namias N, Doherty J, Manning RJ, Li P, Elhaddad A, Lasko D, Amortegui J, Dy CJ, Dlugasch L, Baracco G, Cohn SM. The effect of antipyretic therapy upon outcomes in critically ill patients: a randomized, prospective study. Surg Infect (Larchmt). 2005 Winter;6(4):369-75. doi: 10.1089/sur.2005.6.369. PMID 16433601
- [Background] Young P, Saxena M, Bellomo R, Freebairn R, Hammond N, van Haren F, Holliday M, Henderson S, Mackle D, McArthur C, McGuinness S, Myburgh J, Weatherall M, Webb S, Beasley R; HEAT Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Acetaminophen for Fever in Critically Ill Patients with Suspected Infection. N Engl J Med. 2015 Dec 3;373(23):2215-24. doi: 10.1056/NEJMoa1508375. Epub 2015 Oct 5. PMID 26436473
- [Background] Ye S, Xu D, Zhang C, Li M, Zhang Y. Effect of Antipyretic Therapy on Mortality in Critically Ill Patients with Sepsis Receiving Mechanical Ventilation Treatment. Can Respir J. 2017;2017:3087505. doi: 10.1155/2017/3087505. Epub 2017 Mar 12. PMID 28386165
- [Background] Bernard GR, Wheeler AP, Russell JA, Schein R, Summer WR, Steinberg KP, Fulkerson WJ, Wright PE, Christman BW, Dupont WD, Higgins SB, Swindell BB. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. N Engl J Med. 1997 Mar 27;336(13):912-8. doi: 10.1056/NEJM199703273361303. PMID 9070471